CLINICAL TRIAL: NCT05483647
Title: Erector Spine Plane Block as a Component of General Anesthesia in Spine Surgery
Brief Title: ERECTOR SPINE PLANE BLOCK VERSUS LOCAL INFILTRATION ANAESTHESIA FOR TRANSFORAMINAL PERCUTANEOUS ENDOSCOPIC DISCECTOMY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lviv National Medical University (Other)
Responsible Party: Principal Investigator, Maksym Barsa, Doctor, Lviv National Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LNMY-FPGE- ANESTHESIOLOGY-TPED
Record Dates: First submitted 2022-07-31; First posted 2022-08-02 (Actual); Last update posted 2022-08-04 (Actual); Status verified 2022-08

CONDITIONS: Acute Pain; Chronic Pain; Postoperative Pain; Anesthesia; Regional Anesthesia Morbidity; Anesthesia, Local; Anesthesia Complication; Hyperalgesia; Intraoperative Complications; Intraoperative Neurological Injury; Intraoperative Injury; Postoperative Nausea and Vomiting; Postoperative Cognitive Dysfunction; Neuropathic Pain
Keywords: ERECTOR SPINE PLANE BLOCK; Regional anesthesia; LOCAL INFILTRATION ANAESTHESIA; TRANSFORAMINAL PERCUTANEOUS ENDOSCOPIC DISCECTOMY
MeSH Terms: conditions — Acute Pain; Chronic Pain; Pain, Postoperative; Hyperalgesia; Intraoperative Complications; Postoperative Nausea and Vomiting; Postoperative Cognitive Complications; Neuralgia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- G1 (Active Comparator): Intravenous sedation with infiltrative local anaesthesia
  Interventions: Procedure: Local infiltrative anaesthesia
- G2 (Experimental): Intravenous sedation with bilateral Erector Spine Plane Block
  Interventions: Procedure: Erector spine plane block

INTERVENTIONS:
Procedure: Local infiltrative anaesthesia — In prone position, before the skin incision, patients in G1 underwent local infiltrative anaesthesia et the level of incision. The skin, subcutaneous tissue and muscles up to the foramen intervertebral were anesthetized by the surgeon employing forty millilitre solution of Lidocaine 1% with Dexamethasone 0.02% and Epinephrine 0.00018%.
  Arms: G1
Procedure: Erector spine plane block — The transverse vertebral process of the required level of spine was identified using the mobile C-arm X-ray System. When the tip of the 22G needle reached to the transverse vertebral process 3 cm lateral to the spinous process, a solution of 40 millilitres of Lidocaine 1% with Dexamethasone 0.02% and Epinephrine 0.00018% was injected under the erector spinae muscle bilaterally.
  Arms: G2

SUMMARY:
The main aim of our study was to test the hypothesis that Erector spine plane block (ESP) with sedation will provide the similar employment of fentanyl and propofol during surgery as an infiltrative local anaesthesia with sedation. The primary endpoint was the quantity of fentanyl and propofol during surgery.

DETAILED DESCRIPTION:
Primary outcome: amount of fentanyl and propofol during surgery. Secondary outcomes: adverse events during sedation using World Society of Intravenous Anaesthesia (SIVA) adverse sedation event reporting tool [15], level of postoperative sedation with Richmond Agitation-Sedation Scale (RASS), intensity of pain after surgery using a visual analogue scale (VAS), the mechanical pain threshold (MPT) with von Frey monofilaments measured on both lower extremities, satisfaction with analgesia using 5-point Likert scale.

In both groups, intraoperative analgesia was provided by fentanyl, intraoperative sedation by propofol. Fentanyl was administered to the patients of booth groups in the case of low back pain complaint and/or increasing in heart rate and blood pressure more than 20% of baseline in the dose of 50 μg. If case of sharp shooting pain in lower extremity the surgeon changed the position of the endoscope in order not to irritate the spinal cord root, fentanyl was not administrated.

After performing the local infiltrative anaesthesia or ESP, propofol was given by target-controlled infusion based on the propofol pharmacokinetic parameters reported by Eleveld 2.1 [16]. The initial propofol plasma concentration target was 1,0 μg ml-1 in both groups (we used iTIVA plus Anaesthesia software v5.2.3 to predict the propofol concentrations). Subsequently, the infusion rate of propofol was changed in order to reach not less than 2-3 score levels of modified observer's assessment of alertness/sedation scale (MOAA/S).

During procedural sedation was used World SIVA adverse sedation event reporting tool. All five steps which require this tool were completed. If there were one or more adverse events associated with this sedation encounter (minimal risk descriptors, minor risk descriptors, sentinel risk descriptors or other) they were described. Interventions that were performed to treat the adverse events and the outcomes of the adverse events were also noted.

After the discharge from the operating room to postoperative ward, the level of postoperative sedation was accessed using RASS. Two hours after surgery intensity of pain and the mechanical pain threshold were obtained as well as satisfaction with analgesia using 5-point Likert scale.

To determine the mechanical pain threshold after surgery Von Frey monofilaments were used. The set consists of 20 nylon filaments of different thicknesses in ascending order. Patients were asked to lie down on their backs, close their eyes and inform the doctor when they felt a clear point of contact with the skin. Monofilaments were pressed against the skin of the middle third of the palmar surface of the forearm at an angle of 90 ° until the filament bends for 2 seconds. Monofilaments were used in ascending order with an interval of 10 seconds.

All patients in the operating room received paracetamol, dexketoprofen, ondansetron, dexamethasone, and tranexamic acid. In prone position, before the skin incision, patients in G1 underwent local infiltrative anaesthesia et the level of incision. The skin, subcutaneous tissue and muscles up to the foramen intervertebral were anesthetized by the surgeon employing forty millilitre solution of Lidocaine 1% with Dexamethasone 0.02% and Epinephrine 0.00018%. Patients in G2 underwent bilateral ESP. The transverse vertebral process of the required level of spine was identified using the mobile C-arm X-ray System. When the tip of the 22G needle reached to the transverse vertebral process 3 cm lateral to the spinous process, a solution of 40 millilitres of Lidocaine 1% with Dexamethasone 0.02% and Epinephrine 0.00018% was injected under the erector spinae muscle bilaterally. For postoperative analgesia, patients in both groups received nonsteroidal anti-inflammatory drugs (paracetamol in combination with dexketoprofen) every six hours. Thromboprophylaxis was administered based on the risk of thromboembolic complications.

Duration of observation of the patients was proceed until discharge from the hospital.

ELIGIBILITY:
Inclusion Criteria: informed consent of the patient to participate in the study, intervertebral hernia that require transforaminal percutaneous endoscopic discectomy, and the absence of known allergies to local anaesthetics.

Exclusion Criteria: refusal to participate in the study both at the beginning of the study and at any stage of the study, physical status according to the ASA classification III and more, age more than 50 years old, body mass index (BMI) more than 30 kg/m2.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-07-05 (Actual)

PRIMARY OUTCOMES:
Amount of fentanyl and propofol during surgery | Through study completion, an average of 1 year

SECONDARY OUTCOMES:
Adverse events during sedation using World Society of Intravenous Anaesthesia adverse sedation event reporting tool | Through study completion, an average of 1 year
Level of postoperative sedation with Richmond Agitation-Sedation Scale | Through study completion, an average of 1 year
Intensity of pain after surgery using a visual analogue scale | On hour after surgery
The mechanical pain threshold with von Frey monofilaments measured on both lower extremities | Baseline, on the 1st day after surgery
Satisfaction with analgesia using 5-point Likert scale. | On the 5st day after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Rivne Oblast State Hospital, Rivne, Rivne Oblast, Ukraine

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP